CLINICAL TRIAL: NCT01295827
Title: Phase I Study of Single Agent Pembrolizumab (MK-3475) in Patients With Progressive Locally Advanced or Metastatic Carcinoma, Melanoma, and Non-Small Cell Lung Carcinoma (KEYNOTE 001)
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Progressive Locally Advanced or Metastatic Carcinoma, Melanoma, or Non-small Cell Lung Carcinoma (P07990/MK-3475-001/KEYNOTE-001)
Acronym: KEYNOTE-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07990; MK-3475-001 (Other: Merck Protocol Number); 2011-002371-42 (EudraCT Number); P07990 (Other: Merck); KEYNOTE-001 (Other: Merck)
Record Dates: First submitted 2011-02-10; First posted 2011-02-15 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Cancer, Solid Tumor
Keywords: Melanoma; Carcinoma; Cancer; Advanced cancer; Metastatic cancer; Metastatic melanoma; Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma; Neoplasm Metastasis; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) (Experimental): During Cycle 1 participants received a dose of 1 mg/kg pembrolizumab intravenous (IV) infusion over 30 minutes on Day 1 of a 28-day cycle for evaluation of dose-limiting toxicities and pharmacokinetics. Participants received pembrolizumab IV at a dose of 1 mg/kg every 2 weeks (Q2W) starting with Cycle 2.
  Interventions: Biological: Pembrolizumab
- Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) (Experimental): During Cycle 1 participants received a dose of 3 mg/kg pembrolizumab IV infusion over 30 minutes on Day 1 of a 28-day cycle for evaluation of dose-limiting toxicities and pharmacokinetics. Participants received pembrolizumab IV at a dose of 3 mg/kg Q2W starting with Cycle 2.
  Interventions: Biological: Pembrolizumab
- Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) (Experimental): During Cycle 1 participants received a dose of 10 mg/kg pembrolizumab IV infusion over 30 minutes on Day 1 of a 28-day cycle for evaluation of dose-limiting toxicities and pharmacokinetics. Participants received pembrolizumab IV at a dose of 10 mg/kg Q2W starting with Cycle 2.
  Interventions: Biological: Pembrolizumab
- Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) (Experimental): During Cycle 1 participants received pembrolizumab dose titration from 0.005 mg/kg to 0.3 mg/kg to 2.0 mg/kg on Days 1, 8, and 22, administered as an IV infusion over 30 minutes. Participants received 2 mg/kg every 3 weeks (Q3W) starting with Cycle 2.
  Interventions: Biological: Pembrolizumab
- Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) (Experimental): During Cycle 1 participants received pembrolizumab dose titration from 0.02 mg/kg to 0.3 mg/kg to 2.0 mg/kg on Days 1, 8, and 22, administered as an IV infusion over 30 minutes. Participants received 2 mg/kg Q3W starting with Cycle 2.
  Interventions: Biological: Pembrolizumab
- Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) (Experimental): During Cycle 1 participants received pembrolizumab dose titration from 0.06 mg/kg to 1.0 mg/kg to 10 mg/kg on Days 1, 8, and 22, administered as an IV infusion over 30 minutes. Participants received 10 mg/kg Q3W starting with Cycle 2.
  Interventions: Biological: Pembrolizumab
- MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) (Experimental): Participants received pembrolizumab IV at a dose of 2 mg/kg Q2W. After Amendment 3, participants received dosing Q3W. After Amendment 10, all remaining and ongoing participants were treated with a 200 mg fixed dose of pembrolizumab IV Q3W based on analysis of safety and efficacy data.
  Interventions: Biological: Pembrolizumab
- MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) (Experimental): Participants received pembrolizumab IV at a dose of 10 mg/kg Q2W. After Amendment 7, participants received dosing Q3W. After Amendment 10, all remaining and ongoing participants were treated with a 200 mg fixed dose of pembrolizumab IV Q3W based on analysis of safety and efficacy data.
  Interventions: Biological: Pembrolizumab
- MEL: Pembrolizumab 10 mg/kg Q2W (Part B) (Experimental): Participants received pembrolizumab IV at a dose of 10 mg/kg Q2W. After Amendment 10, all remaining and ongoing participants were treated with a 200 mg fixed dose of pembrolizumab IV Q3W based on analysis of safety and efficacy data.
  Interventions: Biological: Pembrolizumab
- NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) (Experimental): Participants received pembrolizumab IV at a dose of 2 mg/kg Q3W. After Amendment 10, all remaining and ongoing participants were treated with a 200 mg fixed dose of pembrolizumab IV Q3W based on analysis of safety and efficacy data.
  Interventions: Biological: Pembrolizumab
- NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) (Experimental): Participants received pembrolizumab IV at a dose of 10 mg/kg Q3W. After Amendment 10, all remaining and ongoing participants were treated with a 200 mg fixed dose of pembrolizumab IV Q3W based on analysis of safety and efficacy data.
  Interventions: Biological: Pembrolizumab
- NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F) (Experimental): Participants received pembrolizumab IV at a dose of 10 mg/kg Q2W. After Amendment 10, all remaining and ongoing participants were treated with a 200 mg fixed dose of pembrolizumab IV Q3W based on analysis of safety and efficacy data.
  Interventions: Biological: Pembrolizumab
- NSCLC: Pembrolizumab 2 mg/kg Q3W (Part E-Not Enrolled) (Experimental): Participants were to receive pembrolizumab IV at a dose of 2 mg/kg Q3W. No participants were enrolled in this arm.
  Interventions: Biological: Pembrolizumab
- NSCLC: Pembrolizumab 5 mg/kg Q3W (Part E-Not Enrolled) (Experimental): Participants were to receive pembrolizumab IV at a dose of 5 mg/kg Q3W. No participants were enrolled in this arm.
  Interventions: Biological: Pembrolizumab
- NSCLC: Pembrolizumab 10 mg/kg Q3W (Part E-Not Enrolled) (Experimental): Participants were to receive pembrolizumab IV at a dose of 10 mg/kg Q3W. No participants were enrolled in this arm.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion over 30 minutes on Day 1 of each cycle, administered according to dose selection or randomization.
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
The present study has 5 parts. In Parts A and A1, the dose of intravenous (IV) pembrolizumab (MK-3475) will be escalated from 1 to 10 mg/kg to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) for participants with a histologically- or cytologically-confirmed diagnosis of any type of carcinoma or melanoma (MEL) by evaluating the Dose Limiting Toxicities (DLTs). Following completion of the dose escalation, additional patients will be enrolled in Part A2 to further define pharmacokinetic characteristics. Part B of the study will investigate the safety, tolerability, and efficacy of pembrolizumab (2 mg/kg and 10 mg/kg) in participants with advanced or metastatic MEL and compare every 2 week dosing (Q2W) to every 3 week dosing (Q3W). Part C of the study will investigate the safety, tolerability, and efficacy of pembrolizumab administered at 10 mg/kg Q3W in participants with non-small cell lung carcinoma (NSCLC) that is locally advanced or metastatic. Part D of the study will investigate the low and high doses of study drug identified in Parts A and B (2 mg/kg and 10 mg/kg) administered Q3W in participants with advanced or metastatic MEL. Part E (closed with Amendment 7) was planned to investigate low, medium, and high doses of pembrolizumab in combination with standard chemotherapy in participants with locally advanced or metastatic NSCLC. Part F will investigate low and high doses of pembrolizumab (2 mg/kg and 10 mg/kg) administered Q2W or Q3W in treatment-naive and previously-treated participants with NSCLC with programmed cell death 1 ligand (PD-L1) gene expression. The primary hypotheses are the following: that pembrolizumab will have acceptable safety and tolerability; that pembrolizumab will show a clinically meaningful response rate (RR) or disease-control rate (DCR) in participants with melanoma (ipilimumab-refractory or not) and NSCLC, and that pembrolizumab will show a more clinically meaningful RR in participants with either cancer whose tumors express PD-L1.

DETAILED DESCRIPTION:
Per protocol, all participants who were receiving study intervention or in survival follow-up could enroll in the extension study, KEYNOTE-587 (NCT03486873), which would allow further study participation after the Primary Completion Date cut-off. Thus, all efficacy outcome measures except for survival (Overall Survival [OS]) were to be followed up to the Interim Database cut-off of 18-Sept-2018, and the primary safety analyses (except for the DLT analysis) and Overall Survival were to be followed up to the study Primary Completion Date (Final Database cut-off of 05-Nov-2018).

Five participants did not have end of study assessments completed by the Primary Completion Date cut-off and were subsequently followed up to the Study Completion Date (11-Dec-2018). End of treatment and end of study assessments are missing for these 5 and the status was noted as unknown as of the Primary Completion Date cut-off. Per protocol, any safety information after the Primary Completion Date cut-off (Final Database cut-off of 05-Nov-2018) would not be included in the safety analysis but reported by the Investigator to the Sponsor via the Sponsor Communication Form and filed in the electronic Trial Master File.

ELIGIBILITY:
Inclusion Criteria

* In Part A: Histological or cytological diagnosis of MEL or any type of carcinoma, progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy. In Parts B and D of the study, histological or cytological diagnoses of metastatic MEL with progressive locally advanced or metastatic disease. In Parts C and F, histological or cytological diagnosis of NSCLC. In Part F1, participants with Stage IV NSCLC without prior systemic therapy may be eligible.
* Failure of established standard medical anti-cancer therapies for a given tumor type or intolerance to such therapy.
* In Parts B, C, D, or F of the study, MEL or NSCLC must be measurable by imaging.
* In Part F of the study, NSCLC with PD-L1 gene expression.
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Adequate organ function.
* Female participants of childbearing potential should have a negative urine or serum pregnancy test prior to receiving study medication
* Female participants of childbearing potential must be willing to use adequate contraception from study start, through the course of the study, and for 120 days after the last dose of study medication
* Male participants of childbearing potential must agree to use adequate contraception from the first dose of study medication through 120 days after the last dose of study medication

Exclusion Criteria

* Chemotherapy, radioactive, or biological cancer therapy within 4 weeks prior to the first dose of study therapy, or not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from the adverse events caused by therapy administered more than 4 weeks prior to first dose.
* Participation in a study of an investigational agent or using an investigational device within 30 days of administration of pembrolizumab, with the exception of participants in the follow-up phase.
* Other form(s) of antineoplastic therapy anticipated during the period of the study.
* History of non-infectious pneumonitis requiring treatment with steroids, or has a history of interstitial lung disease.
* Medical condition that requires chronic systemic steroid therapy, or on any other form of immunosuppressive medication, excepting use of inhaled steroids.
* Risk factors for bowel obstruction or bowel perforation (including a history of acute diverticulitis, intra-abdominal abscess, abdominal carcinomatosis).
* History of a hematologic malignancy, malignant primary brain tumor, malignant sarcoma, or another malignant primary solid tumor, unless no evidence of that disease for 5 years.
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Previous severe hypersensitivity reaction to another monoclonal antibody (mAb).
* Active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents, except vitiligo or resolved childhood asthma/atopy.
* Prior therapy with another anti-programmed cell death (PD)-1 agent or previously enrolled in any pembrolizumab trial.
* Active infection requiring therapy.
* Positive for Human Immunodeficiency Virus (HIV), Hepatitis B (Hepatitis B Surface Antigen [HBsAg] reactive), or Hepatitis C virus (Hepatitis C Virus Ribonucleic Acid [HCV RNA] (qualitative) is detected).
* Regular use of illicit drugs or a recent history (within the last year) of substance abuse (including alcohol).
* Symptomatic ascites or pleural effusion.
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Actual)
Dates: Start 2011-03-04 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Robert C, Ribas A, Wolchok JD, Hodi FS, Hamid O, Kefford R, Weber JS, Joshua AM, Hwu WJ, Gangadhar TC, Patnaik A, Dronca R, Zarour H, Joseph RW, Boasberg P, Chmielowski B, Mateus C, Postow MA, Gergich K, Elassaiss-Schaap J, Li XN, Iannone R, Ebbinghaus SW, Kang SP, Daud A. Anti-programmed-death-receptor-1 treatment with pembrolizumab in ipilimumab-refractory advanced melanoma: a randomised dose-comparison cohort of a phase 1 trial. Lancet. 2014 Sep 20;384(9948):1109-17. doi: 10.1016/S0140-6736(14)60958-2. Epub 2014 Jul 15. PMID 25034862
- [Result] Patnaik A, Kang SP, Rasco D, Papadopoulos KP, Elassaiss-Schaap J, Beeram M, Drengler R, Chen C, Smith L, Espino G, Gergich K, Delgado L, Daud A, Lindia JA, Li XN, Pierce RH, Yearley JH, Wu D, Laterza O, Lehnert M, Iannone R, Tolcher AW. Phase I Study of Pembrolizumab (MK-3475; Anti-PD-1 Monoclonal Antibody) in Patients with Advanced Solid Tumors. Clin Cancer Res. 2015 Oct 1;21(19):4286-93. doi: 10.1158/1078-0432.CCR-14-2607. Epub 2015 May 14. PMID 25977344
- [Result] Chatterjee M, Turner DC, Felip E, Lena H, Cappuzzo F, Horn L, Garon EB, Hui R, Arkenau HT, Gubens MA, Hellmann MD, Dong D, Li C, Mayawala K, Freshwater T, Ahamadi M, Stone J, Lubiniecki GM, Zhang J, Im E, De Alwis DP, Kondic AG, Flotten O. Systematic evaluation of pembrolizumab dosing in patients with advanced non-small-cell lung cancer. Ann Oncol. 2016 Jul;27(7):1291-8. doi: 10.1093/annonc/mdw174. Epub 2016 Apr 26. PMID 27117531
- [Derived] Topp BG, Channavazzala M, Mayawala K, De Alwis DP, Rubin E, Snyder A, Wolchok JD, Ribas A. Tumor dynamics in patients with solid tumors treated with pembrolizumab beyond disease progression. Cancer Cell. 2023 Sep 11;41(9):1680-1688.e2. doi: 10.1016/j.ccell.2023.08.004. PMID 37699333
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] Hamid O, Robert C, Daud A, Carlino MS, Mitchell TC, Hersey P, Schachter J, Long GV, Hodi FS, Wolchok JD, Arance A, Grob JJ, Joshua AM, Weber JS, Mortier L, Jensen E, Diede SJ, Moreno BH, Ribas A. Long-term outcomes in patients with advanced melanoma who had initial stable disease with pembrolizumab in KEYNOTE-001 and KEYNOTE-006. Eur J Cancer. 2021 Nov;157:391-402. doi: 10.1016/j.ejca.2021.08.013. Epub 2021 Sep 25. PMID 34571336
- [Derived] Robert C, Hwu WJ, Hamid O, Ribas A, Weber JS, Daud AI, Hodi FS, Wolchok JD, Mitchell TC, Hersey P, Dronca R, Joseph RW, Boutros C, Min L, Long GV, Schachter J, Puzanov I, Dummer R, Lin J, Ibrahim N, Diede SJ, Carlino MS, Joshua AM. Long-term safety of pembrolizumab monotherapy and relationship with clinical outcome: A landmark analysis in patients with advanced melanoma. Eur J Cancer. 2021 Feb;144:182-191. doi: 10.1016/j.ejca.2020.11.010. Epub 2020 Dec 24. PMID 33360855
- [Derived] Lala M, Li TR, de Alwis DP, Sinha V, Mayawala K, Yamamoto N, Siu LL, Chartash E, Aboshady H, Jain L. A six-weekly dosing schedule for pembrolizumab in patients with cancer based on evaluation using modelling and simulation. Eur J Cancer. 2020 May;131:68-75. doi: 10.1016/j.ejca.2020.02.016. Epub 2020 Apr 15. PMID 32305010
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Garon EB, Hellmann MD, Rizvi NA, Carcereny E, Leighl NB, Ahn MJ, Eder JP, Balmanoukian AS, Aggarwal C, Horn L, Patnaik A, Gubens M, Ramalingam SS, Felip E, Goldman JW, Scalzo C, Jensen E, Kush DA, Hui R. Five-Year Overall Survival for Patients With Advanced Non-Small-Cell Lung Cancer Treated With Pembrolizumab: Results From the Phase I KEYNOTE-001 Study. J Clin Oncol. 2019 Oct 1;37(28):2518-2527. doi: 10.1200/JCO.19.00934. Epub 2019 Jun 2. PMID 31154919
- [Derived] Leighl NB, Hellmann MD, Hui R, Carcereny E, Felip E, Ahn MJ, Eder JP, Balmanoukian AS, Aggarwal C, Horn L, Patnaik A, Gubens M, Ramalingam SS, Lubiniecki GM, Zhang J, Piperdi B, Garon EB. Pembrolizumab in patients with advanced non-small-cell lung cancer (KEYNOTE-001): 3-year results from an open-label, phase 1 study. Lancet Respir Med. 2019 Apr;7(4):347-357. doi: 10.1016/S2213-2600(18)30500-9. Epub 2019 Mar 12. PMID 30876831
- [Derived] Wang M, Chen C, Jemielita T, Anderson J, Li XN, Hu C, Kang SP, Ibrahim N, Ebbinghaus S. Are tumor size changes predictive of survival for checkpoint blockade based immunotherapy in metastatic melanoma? J Immunother Cancer. 2019 Feb 8;7(1):39. doi: 10.1186/s40425-019-0513-4. PMID 30736858
- [Derived] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph R, Weber JS, Dronca R, Mitchell TC, Patnaik A, Zarour HM, Joshua AM, Zhao Q, Jensen E, Ahsan S, Ibrahim N, Ribas A. Five-year survival outcomes for patients with advanced melanoma treated with pembrolizumab in KEYNOTE-001. Ann Oncol. 2019 Apr 1;30(4):582-588. doi: 10.1093/annonc/mdz011. PMID 30715153
- [Derived] Hamid O, Robert C, Ribas A, Hodi FS, Walpole E, Daud A, Arance AS, Brown E, Hoeller C, Mortier L, Schachter J, Long J, Ebbinghaus S, Ibrahim N, Butler M. Antitumour activity of pembrolizumab in advanced mucosal melanoma: a post-hoc analysis of KEYNOTE-001, 002, 006. Br J Cancer. 2018 Sep;119(6):670-674. doi: 10.1038/s41416-018-0207-6. Epub 2018 Sep 11. PMID 30202085
- [Derived] Joseph RW, Elassaiss-Schaap J, Kefford R, Hwu WJ, Wolchok JD, Joshua AM, Ribas A, Hodi FS, Hamid O, Robert C, Daud A, Dronca R, Hersey P, Weber JS, Patnaik A, de Alwis DP, Perrone A, Zhang J, Kang SP, Ebbinghaus S, Anderson KM, Gangadhar TC. Baseline Tumor Size Is an Independent Prognostic Factor for Overall Survival in Patients with Melanoma Treated with Pembrolizumab. Clin Cancer Res. 2018 Oct 15;24(20):4960-4967. doi: 10.1158/1078-0432.CCR-17-2386. Epub 2018 Apr 23. PMID 29685882
- [Derived] Brogden KA, Parashar D, Hallier AR, Braun T, Qian F, Rizvi NA, Bossler AD, Milhem MM, Chan TA, Abbasi T, Vali S. Genomics of NSCLC patients both affirm PD-L1 expression and predict their clinical responses to anti-PD-1 immunotherapy. BMC Cancer. 2018 Feb 27;18(1):225. doi: 10.1186/s12885-018-4134-y. PMID 29486723
- [Derived] Robert C, Ribas A, Hamid O, Daud A, Wolchok JD, Joshua AM, Hwu WJ, Weber JS, Gangadhar TC, Joseph RW, Dronca R, Patnaik A, Zarour H, Kefford R, Hersey P, Zhang J, Anderson J, Diede SJ, Ebbinghaus S, Hodi FS. Durable Complete Response After Discontinuation of Pembrolizumab in Patients With Metastatic Melanoma. J Clin Oncol. 2018 Jun 10;36(17):1668-1674. doi: 10.1200/JCO.2017.75.6270. Epub 2017 Dec 28. PMID 29283791
- [Derived] Shaverdian N, Lisberg AE, Bornazyan K, Veruttipong D, Goldman JW, Formenti SC, Garon EB, Lee P. Previous radiotherapy and the clinical activity and toxicity of pembrolizumab in the treatment of non-small-cell lung cancer: a secondary analysis of the KEYNOTE-001 phase 1 trial. Lancet Oncol. 2017 Jul;18(7):895-903. doi: 10.1016/S1470-2045(17)30380-7. Epub 2017 May 24. PMID 28551359
- [Derived] Hui R, Garon EB, Goldman JW, Leighl NB, Hellmann MD, Patnaik A, Gandhi L, Eder JP, Ahn MJ, Horn L, Felip E, Carcereny E, Rangwala R, Lubiniecki GM, Zhang J, Emancipator K, Roach C, Rizvi NA. Pembrolizumab as first-line therapy for patients with PD-L1-positive advanced non-small cell lung cancer: a phase 1 trial. Ann Oncol. 2017 Apr 1;28(4):874-881. doi: 10.1093/annonc/mdx008. PMID 28168303
- [Derived] Daud AI, Wolchok JD, Robert C, Hwu WJ, Weber JS, Ribas A, Hodi FS, Joshua AM, Kefford R, Hersey P, Joseph R, Gangadhar TC, Dronca R, Patnaik A, Zarour H, Roach C, Toland G, Lunceford JK, Li XN, Emancipator K, Dolled-Filhart M, Kang SP, Ebbinghaus S, Hamid O. Programmed Death-Ligand 1 Expression and Response to the Anti-Programmed Death 1 Antibody Pembrolizumab in Melanoma. J Clin Oncol. 2016 Dec;34(34):4102-4109. doi: 10.1200/JCO.2016.67.2477. Epub 2016 Oct 31. PMID 27863197
- [Derived] Ribas A, Hamid O, Daud A, Hodi FS, Wolchok JD, Kefford R, Joshua AM, Patnaik A, Hwu WJ, Weber JS, Gangadhar TC, Hersey P, Dronca R, Joseph RW, Zarour H, Chmielowski B, Lawrence DP, Algazi A, Rizvi NA, Hoffner B, Mateus C, Gergich K, Lindia JA, Giannotti M, Li XN, Ebbinghaus S, Kang SP, Robert C. Association of Pembrolizumab With Tumor Response and Survival Among Patients With Advanced Melanoma. JAMA. 2016 Apr 19;315(15):1600-9. doi: 10.1001/jama.2016.4059. PMID 27092830
- [Derived] Hodi FS, Hwu WJ, Kefford R, Weber JS, Daud A, Hamid O, Patnaik A, Ribas A, Robert C, Gangadhar TC, Joshua AM, Hersey P, Dronca R, Joseph R, Hille D, Xue D, Li XN, Kang SP, Ebbinghaus S, Perrone A, Wolchok JD. Evaluation of Immune-Related Response Criteria and RECIST v1.1 in Patients With Advanced Melanoma Treated With Pembrolizumab. J Clin Oncol. 2016 May 1;34(13):1510-7. doi: 10.1200/JCO.2015.64.0391. Epub 2016 Mar 7. PMID 26951310
- [Derived] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Derived] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph RW, Weber JS, Dronca R, Gangadhar TC, Patnaik A, Zarour H, Joshua AM, Gergich K, Elassaiss-Schaap J, Algazi A, Mateus C, Boasberg P, Tumeh PC, Chmielowski B, Ebbinghaus SW, Li XN, Kang SP, Ribas A. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma. N Engl J Med. 2013 Jul 11;369(2):134-44. doi: 10.1056/NEJMoa1305133. Epub 2013 Jun 2. PMID 23724846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a histologically- or cytologically-confirmed diagnosis of any type of carcinoma (solid tumors), melanoma (MEL), or non-small cell lung cancer (NSCLC), with progressive locally advanced or metastatic disease, were recruited.
Pre-assignment Details: Of 1260 participants enrolled or randomized to the study, 1235 received at least one dose of treatment (All Treated Population) and were evaluable for all safety and efficacy analyses. Part E did not enroll any participants.
Period: Overall Study
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part E-Not Enrolled) | NSCLC: Pembrolizumab 5 mg/kg Q3W (Part E-Not Enrolled) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Part E-Not Enrolled)
Started | 4 | 3 | 12 | 4 | 3 | 6 | 164 | 321 | 183 | 61 | 296 | 203 | 0 | 0 | 0
Treated (All Treated Population) | 4 | 3 | 10 | 4 | 3 | 6 | 162 | 313 | 180 | 61 | 287 | 202 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 18 | 24 | 14 | 6 | 20 | 17 | 0 | 0 | 0
Not Completed | 4 | 3 | 12 | 4 | 2 | 6 | 146 | 297 | 169 | 55 | 276 | 186 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 2 | 1 | 1 | 4 | 15 | 49 | 22 | 7 | 50 | 21 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 1 | 0 | 4 | 8 | 7 | 4 | 7 | 3 | 0 | 0 | 0
Not completed — Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 24 | 58 | 41 | 2 | 23 | 13 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 1 | 5 | 2 | 0 | 1 | 87 | 144 | 85 | 40 | 175 | 136 | 0 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0 | 0 | 1 | 13 | 35 | 11 | 2 | 18 | 13 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A): During Cycle 1 participants received a dose of 1 mg/kg pembrolizumab IV infusion over 30 minutes on Day 1 of a 28-day cycle for evaluation of dose-limiting toxicities and pharmacokinetics. Participants received pembrolizumab IV at a dose of 1 mg/kg Q2W starting with Cycle 2.
- Total: Total of all reporting groups
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F) | Total
Number analyzed (Participants) | 4 | 3 | 12 | 4 | 3 | 6 | 164 | 321 | 183 | 61 | 296 | 203 | 1260
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.0 (6.4) | 76.0 (8.7) | 62.7 (16.1) | 53.8 (11.7) | 53.3 (23.5) | 69.0 (7.6) | 57.9 (13.5) | 60.5 (13.5) | 60.1 (14.4) | 61.9 (11.0) | 61.8 (11.2) | 63.0 (10.2) | 61.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 0 | 0 | 0 | 69 | 125 | 122 | 29 | 145 | 91 | 589
  Male | 1 | 1 | 9 | 4 | 3 | 6 | 95 | 196 | 61 | 32 | 151 | 112 | 671
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3 | 0 | 0 | 0 | 12 | 13 | 3 | 1 | 20 | 8 | 63
  Not Hispanic or Latino | 2 | 2 | 9 | 4 | 3 | 6 | 152 | 308 | 180 | 60 | 274 | 195 | 1195
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 2 | 6 | 46 | 19 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 12 | 8 | 26
  White | 4 | 3 | 12 | 4 | 2 | 6 | 161 | 310 | 178 | 53 | 237 | 174 | 1144
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v.4.0) in Participants With Solid Tumors (Parts A and A1)
Description: DLTs were assessed according to NCI-CTCAE v.4.0 during the first cycle (28 days) and were defined as occurrence of any of the following toxicities if judged by the investigator to be possibly, probably or definitely related to study drug administration: Grade (Gr) 4 nonhematologic toxicity; Gr 4 hematologic toxicity lasting ≥14 days; Gr 3 nonhematologic toxicity lasting >3 days despite optimal supportive care; any Grade 3 non-hematologic laboratory value if medical intervention was required to treat the participant, the abnormality led to hospitalization, or the abnormality persisted for >1 week; Gr 3 or 4 febrile neutropenia; thrombocytopenia <25,000 cells/mm^3 (if associated with a bleeding event requiring an elective platelet transfusion, or a life-threatening bleeding event which resulted in urgent intervention and admission to an Intensive Care Unit); or Gr 5 toxicity. The number of participants in Part A and Part A1 with a DLT were reported by pembrolizumab dose received.
Time Frame: Up to 28 days in Cycle 1
Population: All participants in Parts A and A1 who received ≥1 dose of study treatment and either 1) had a DLT in Cycle 1 or 2) received ≥90% of the prescribed dose of pembrolizumab in Cycle 1 and completed all safety evaluations ≥28 days after the first administration of pembrolizumab without experiencing DLT. Per protocol, Parts A2 and B-F were not analyzed.
Measure: Number; unit: Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 4 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 0 |  |  |  |  |  |  |  |  |

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which was temporally associated with the use of the Sponsor's product was also an AE. The number of participants who experienced an AE was reported for each arm.
Time Frame: Up to approximately 91 months (through Final Database cut-off date of 05-Nov-2018)
Population: All participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 4 | 3 | 10 | 4 | 3 | 6 | 162 | 313 | 180 | 61 | 287 | 202
Participants | 4 | 3 | 9 | 4 | 3 | 6 | 161 | 308 | 178 | 60 | 277 | 198

3. Primary Outcome: Overall Response Rate (ORR) According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Integrated Radiology and Oncology (IRO): Melanoma Participants (Parts B Plus D)
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR: disappearance of all lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) according to RECIST 1.1, which was modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a confirmed CR or PR according to RECIST 1.1 as assessed by IRO was reported as the ORR for each melanoma dose arm (Parts B plus D).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: All melanoma (Parts B plus D) participants that received ≥1 dose of study treatment. Per protocol, Part A (dose-escalation) was not analyzed for efficacy. NSCLC (Parts C plus F) participants were analyzed and presented separately and are not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 162 | 313 | 180 | 0 | 0 | 0
Percentage of Participants |  |  |  |  |  |  | 30.2 [23.3 to 37.9] | 29.4 [24.4 to 34.8] | 36.7 [29.6 to 44.2] |  |  |

4. Primary Outcome: ORR According to RECIST 1.1 as Assessed by Independent Review Committee (IRC): Non-Small Cell Lung Cancer (NSCLC) Participants (Parts C Plus F)
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed CR (disappearance of all lesions) or PR (at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) according to RECIST 1.1, which was modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a confirmed CR or PR according to RECIST 1.1 as assessed by IRC was reported as the ORR for each NSCLC dose arm (Parts C plus F).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: All NSCLC (Parts C plus F) participants that received ≥1 dose of study treatment. Per protocol, Part A (dose-escalation) was not analyzed for efficacy. Melanoma (Parts B plus D) participants were analyzed and presented separately and are not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 287 | 202
Percentage of Participants |  |  |  |  |  |  |  |  |  | 19.7 [10.6 to 31.8] | 21.6 [17.0 to 26.8] | 19.3 [14.1 to 25.4]

5. Secondary Outcome: ORR According to Immune-related Response Criteria (irRC) as Assessed by Investigator in Melanoma Participants (Parts B Plus D)
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed immune-related Complete Response (irCR: complete disappearance of all tumor lesions whether measurable or not, and no new lesions) or immune-related Partial Response (irPR: decrease in sum of the products of the two largest perpendicular diameters (SPD) of ≥50% by a consecutive assessment ≥4 weeks after first documentation) according to irRC. The percentage of participants who experienced a confirmed irCR or irPR according to irRC as assessed by the investigator was reported as the ORR for each melanoma dose arm (Parts B plus D).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 162 | 313 | 180 | 0 | 0 | 0
Percentage of Participants |  |  |  |  |  |  | 35.2 [27.9 to 43.1] | 39.9 [34.5 to 45.6] | 45.6 [38.1 to 53.1] |  |  |

6. Secondary Outcome: ORR According to irRC as Assessed by Investigator in NSCLC Participants (Parts C Plus F)
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed irCR (complete disappearance of all tumor lesions whether measurable or not, and no new lesions) or irPR (decrease in sum of the products of the two largest perpendicular diameters (SPD) of ≥50% by a consecutive assessment ≥4 weeks after first documentation) according to irRC. The percentage of participants who experienced a confirmed irCR or irPR according to irRC as assessed by the investigator was reported as the ORR for each NSCLC dose arm (Parts C plus F).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 287 | 202
Percentage of Participants |  |  |  |  |  |  |  |  |  | 23.0 [13.2 to 35.5] | 28.9 [23.7 to 34.5] | 22.3 [16.7 to 28.6]

7. Secondary Outcome: Area Under the Concentration-Time Curve of Pembrolizumab From Time 0 to Day 28 (AUC 0-28) in Solid Tumor Participants (Parts A and A1)
Description: Blood samples were collected at specified intervals for the determination of AUC0-28. AUC0-28 was defined as the area under the concentration-time curve of pembrolizumab from time zero to Day 28. AUC0-28 was based on noncompartmental analysis and reported for participants in Parts A and A1.
Time Frame: Cycle 1: Pre-dose, post-dose at 0.5, 6, 24, and 48 hours and Days 8, 15, and 22 (Cycle 1 = 28 days)
Population: All participants in Parts A and A1 receiving a single dose of drug during Cycle 1 (28 days) and having available AUC0-28 data. Two participants were excluded from analysis due to discontinuation. Per protocol, participants in Parts A2, B, C, D, C, and F were not included in the single dose pharmacokinetic (PK) analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg•day/mL
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 3 | 3 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
μg•day/mL | 157 (16) | 955 (23) | 2160 (31) |  |  |  |  |  |  |  |  |

8. Secondary Outcome: Area Under the Concentration-Time Curve of Pembrolizumab From Time 0 to Infinity (AUC 0-inf) in Solid Tumor Participants (Parts A and A1)
Description: Blood samples were collected at specified intervals for the determination of AUC0-inf. AUC0-inf was defined as the area under the concentration-time curve of pembrolizumab from time zero to infinity. AUC0-inf was based on noncompartmental analysis and reported for participants in Parts A and A1.
Time Frame: Cycle 1: Pre-dose, post-dose at 0.5, 6, 24, and 48 hours and Days 8, 15, and 22 (Cycle 1 = 28 days)
Population: All participants in Parts A and A1 receiving a single dose of drug during Cycle 1 (28 days) and having available AUC0-inf data. Two participants were excluded from analysis due to discontinuation. Per protocol, participants in Parts A2, B, C, D, C, and F were not included in the single dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg•day/mL
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 3 | 3 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
μg•day/mL | 212 (36) | 1530 (28) | 3230 (44) |  |  |  |  |  |  |  |  |

9. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab in Solid Tumor Participants (Parts A and A1)
Description: Blood samples were collected at specified intervals for the determination of Cmax. Cmax was defined as the maximum concentration of pembrolizumab reached. Cmax was based on noncompartmental analysis and reported for participants in Parts A and A1.
Time Frame: Cycle 1: Pre-dose, post-dose at 0.5, 6, 24, and 48 hours and Days 8, 15, and 22 (Cycle 1 = 28 days)
Population: All participants in Parts A and A1 receiving a single dose of drug during Cycle 1 (28 days) and having available Cmax data. Per protocol, participants in Parts A2, B, C, D, C, and F were not included in the single dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 4 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
μg/mL | 16.4 (22) | 107 (26) | 256 (37) |  |  |  |  |  |  |  |  |

10. Secondary Outcome: Time to Maximum Concentration (Tmax) of Pembrolizumab in Solid Tumor Participants (Parts A and A1)
Description: Blood samples were collected at specified intervals for the determination of Tmax. Tmax was defined as time to the maximum concentration of pembrolizumab reached. Tmax was based on noncompartmental analysis and reported for participants in Parts A and A1.
Time Frame: Cycle 1: Pre-dose, post-dose at 0.5, 6, 24, and 48 hours and Days 8, 15, and 22 (Cycle 1 = 28 days)
Population: All participants in Parts A and A1 receiving a single dose of drug during Cycle 1 (28 days) and having available Tmax data. Per protocol, participants in Parts A2, B, C, D, C, and F were not included in the single dose PK analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 4 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
days | 0.05 [0.02 to 0.17] | 0.17 [0.17 to 0.17] | 0.17 [0.03 to 0.99] |  |  |  |  |  |  |  |  |

11. Secondary Outcome: Terminal Half-Life (t ½) of Pembrolizumab in Solid Tumor Participants (Parts A and A1)
Description: Blood samples were collected at specified intervals for the determination of t½. t½ was defined as the time required to divide the pembrolizumab plasma concentration by two after reaching pseudo-equilibrium, following a single dose of pembrolizumab. t½ was based on noncompartmental analysis and reported for participants in Parts A and A1.
Time Frame: Cycle 1: Pre-dose, post-dose at 0.5, 6, 24, and 48 hours and Days 8, 15, and 22 (Cycle 1 = 28 days)
Population: All participants in Parts A and A1 receiving a single dose of drug during Cycle 1 (28 days) and having available t½ data. Two participants were excluded from analysis due to discontinuation. Per protocol, participants in Parts A2, B, C, D, C, and F were not included in the single dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 3 | 3 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
days | 14.1 (51) | 21.6 (10) | 17.5 (54) |  |  |  |  |  |  |  |  |

12. Secondary Outcome: Area Under the Concentration-Time Curve of Pembrolizumab From Time 0 to Day 21 (AUC 0-21) in Solid Tumor Participants (Part A2)
Description: Blood samples were collected at specified intervals for the determination of AUC0-21. AUC0-21 was defined as the area under the concentration-time curve of pembrolizumab from time zero to Study Day 21. AUC0-21 was based on noncompartmental analysis and reported for participants in Part A2.
Time Frame: Cycle 1: Day 1: Pre-dose, post-dose at 0.5, 6, 24, and 48 hours; Day 5, Day 8: pre- and post-dose; Day 15 (Cycle = 21 days)
Population: All participants in Part A2 receiving escalating doses of drug during Cycle 1 (21 days) and having available AUC0-21 data. One participant was excluded from analysis due to discontinuation. Per protocol, participants in Parts A, A1, B, C, D, C, and F were not included in the escalating dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg•day/mL
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
μg•day/mL |  |  |  | 57.1 (21) | 50.4 (28) | 186 (28) |  |  |  |  |  |

13. Secondary Outcome: Area Under the Concentration-Time Curve of Pembrolizumab From Day 21 to Day 42 (AUC21-42) in Solid Tumor Participants (Part A2)
Description: Blood samples were collected at specified intervals for the determination of AUC21-42. AUC21-42 was defined as the area under the concentration-time curve of pembrolizumab from Study Day 21 (end of Cycle 1) through Study Day 42 (end of Cycle 2). AUC21-42 was based on noncompartmental analysis and reported for participants in Part A2.
Time Frame: Cycle 1: Day 21; Cycle 2: Day 1: Pre-dose, post-dose at 0.5 and 24 hours, Day 3, Day 8, Day 15 (Cycle = 21 days)
Population: All participants in Part A2 receiving escalating doses of drug during Cycle 1 and having available AUC21-42 data during Cycle 2. Two participants were excluded from analysis due to discontinuation. Per protocol, participants in Parts A, A1, B, C, D, C, and F were not included in the escalating dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg•day/mL
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
μg•day/mL |  |  |  | 486 (16) | 348 (18) | 2280 (24) |  |  |  |  |  |

14. Secondary Outcome: Lowest Plasma Concentration (Ctrough) of Pembrolizumab in Solid Tumor Participants (Parts A, A1, and A2)
Description: Pre-dose samples were collected 24 hours before infusion of pembrolizumab at specified intervals for the determination of Ctrough. Ctrough was defined as the lowest concentration of pembrolizumab reached before the next dose was administered. Ctrough was reported for each Part A arm according to cycle and nominal time after first dose (Day). Results for each cycle reported for arms with N>1 at that timepoint. Ctrough data for melanoma (Parts B and D) and NSCLC (Parts C and F) participants are presented separately and are not included here.
Time Frame: Parts A and A1: pre-dose at Cycles 2, 4, 6, 8, 10, 12, 14 (cycle=14 days); A2 Cohorts: pre-dose at Cycles 2, 3, 5, 7, 9, 11 (cycle=21 days)
Population: All Part A participants receiving ≥1 dose of drug and having available Ctrough samples collected pre-dose before each cycle. Due to differing dosing schedules or N<1, some time points were not applicable for certain arms if data were not collected or analyzed (indicated by zero participants analyzed entered in the table).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2)
Number analyzed (Participants) | 3 | 3 | 8 | 4 | 3 | 5
μg/mL
  Cycle 2 (Day 21): number analyzed (Participants) | 0 | 0 | 0 | 4 | 3 | 5
  Cycle 2 (Day 21) |  |  |  | 2.3 (46.2) | 1.9 (19.9) | 7.77 (46.1)
  Cycle 2 (Day 28): number analyzed (Participants) | 3 | 3 | 8 | 0 | 0 | 0
  Cycle 2 (Day 28) | 2.19 (62.4) | 18.8 (42.1) | 41.7 (44.6) |  |  |
  Cycle 3 (Day 42): number analyzed (Participants) | 0 | 0 | 0 | 4 | 2 | 3
  Cycle 3 (Day 42) |  |  |  | 10.6 (15.9) | 11.1 (28.9) | 70.1 (15.6)
  Cycle 4 (Day 56): number analyzed (Participants) | 2 | 2 | 4 | 0 | 0 | 0
  Cycle 4 (Day 56) | 6.45 (13) | 50.0 (36.9) | 122 (37.2) |  |  |
  Cycle 5 (Day 84): number analyzed (Participants) | 0 | 0 | 0 | 3 | 2 | 3
  Cycle 5 (Day 84) |  |  |  | 14.8 (33.4) | 18.3 (34.1) | 126 (53.9)
  Cycle 6 (Day 84): number analyzed (Participants) | 2 | 2 | 3 | 0 | 0 | 0
  Cycle 6 (Day 84) | 9.93 (5.6) | 55.2 (33.8) | 168 (49.5) |  |  |
  Cycle 8 (Day 112): number analyzed (Participants) | 0 | 2 | 2 | 0 | 0 | 0
  Cycle 8 (Day 112) |  | 66.8 (11.1) | 260 (1.4) |  |  |
  Cycle 7 (Day 126): number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 3
  Cycle 7 (Day 126) |  |  |  | 29.9 (7.3) | 22.1 (49.2) | 151 (48)
  Cycle 10 (Day 140): number analyzed (Participants) | 0 | 2 | 2 | 0 | 0 | 0
  Cycle 10 (Day 140) |  | 63.0 (29.8) | 200 (4.9) |  |  |
  Cycle 9 (Day 168): number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 3
  Cycle 9 (Day 168) |  |  |  | 29.8 (1) |  | 150 (29.4)
  Cycle 12 (Day 168): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0
  Cycle 12 (Day 168) |  | 62.8 (1.7) |  |  |  |
  Cycle 14 (Day 196): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0
  Cycle 14 (Day 196) |  | 54.1 (4.3) |  |  |  |
  Cycle 11 (Day 210): number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 2
  Cycle 11 (Day 210) |  |  |  | 40.7 (38.6) |  | 179 (37.8)

15. Secondary Outcome: Ctrough of Pembrolizumab in Melanoma Participants (Parts B and D)
Description: Pre-dose samples were collected 24 hours before infusion of pembrolizumab at specified intervals for the determination of Ctrough. Ctrough was defined as the lowest concentration of pembrolizumab reached before the next dose was administered. For the purposes of the Ctrough analysis, samples were collected and analyzed separately for each Part B and D enrolment cohort, and Ctrough was reported for each cohort according to cycle and nominal time after first dose (Day). Results for each cycle reported for arms with N>1 at that timepoint. Ctrough data for solid tumor (Part A) and NSCLC (Parts C and F) participants are presented separately and are not included here.
Time Frame: Part B arms treated every 3 weeks: pre-dose at Cycles 2,5,9,13,17,25,33 (cycle=21 days); Part B treated every 2 weeks: pre-dose at Cycles 2,3,7,13,19,25,31,37 (cycle=14 days); Part D: pre-dose at Cycles 2,3,6,8,12,16,24,32 (cycle=21 days)
Population: All melanoma participants receiving ≥1 dose of drug and having available samples collected pre-dose before each cycle. Per protocol, Ctrough analyzed separately by Part, dose, and dosing schedule. Due to differing dosing schedules, some time points were not applicable for certain arms (indicated by zero participants analyzed entered in the table).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- MEL: Pembrolizumab 2 mg/kg Q3W (Part B); MEL: Pembrolizumab 2 mg/kg Q3W (Part D): Participants received pembrolizumab IV at a dose of 2 mg/kg Q3W.
- MEL: Pembrolizumab 10 mg/kg Q3W (Part B); MEL: Pembrolizumab 10 mg/kg Q3W (Part D): Participants received pembrolizumab IV at a dose of 10 mg/kg Q3W.
- MEL: Pembrolizumab 10 mg/kg Q2W (Part B): Participants received pembrolizumab IV at a dose of 10 mg/kg Q2W.
Arm/Group | MEL: Pembrolizumab 2 mg/kg Q3W (Part B) | MEL: Pembrolizumab 10 mg/kg Q3W (Part B) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | MEL: Pembrolizumab 2 mg/kg Q3W (Part D) | MEL: Pembrolizumab 10 mg/kg Q3W (Part D)
Number analyzed (Participants) | 91 | 208 | 150 | 52 | 48
µg/mL
  Cycle 2 (Day 14): number analyzed (Participants) | 0 | 0 | 5 | 0 | 0
  Cycle 2 (Day 14) |  |  | 63.7 (13.6) |  |
  Cycle 2 (Day 21): number analyzed (Participants) | 91 | 208 | 0 | 52 | 48
  Cycle 2 (Day 21) | 8.69 (48.9) | 48.5 (37.9) |  | 10.1 (56.3) | 62.6 (37.2)
  Cycle 3 (Day 28): number analyzed (Participants) | 0 | 0 | 150 | 0 | 0
  Cycle 3 (Day 28) |  |  | 94.0 (47.2) |  |
  Cycle 3 (Day 42): number analyzed (Participants) | 0 | 2 | 0 | 46 | 46
  Cycle 3 (Day 42) |  | 80.3 (1.2) |  | 16.8 (57.2) | 94.3 (37.1)
  Cycle 5 (Day 84): number analyzed (Participants) | 60 | 154 | 0 | 0 | 0
  Cycle 5 (Day 84) | 19.5 (58.3) | 119 (50.7) |  |  |
  Cycle 7 (Day 84): number analyzed (Participants) | 0 | 0 | 110 | 0 | 0
  Cycle 7 (Day 84) |  |  | 173 (49.7) |  |
  Cycle 6 (Day 105): number analyzed (Participants) | 0 | 0 | 0 | 35 | 33
  Cycle 6 (Day 105) |  |  |  | 25.3 (52.4) | 132 (45.6)
  Cycle 7 (Day 126): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Cycle 7 (Day 126) |  | 89.2 (34.4) |  |  |
  Cycle 8 (Day 147): number analyzed (Participants) | 0 | 2 | 0 | 31 | 29
  Cycle 8 (Day 147) |  | 166 (5.1) |  | 23.5 (50.1) | 152 (40.7)
  Cycle 9 (Day 168 ): number analyzed (Participants) | 44 | 112 | 0 | 0 | 0
  Cycle 9 (Day 168 ) | 25.5 (59.6) | 161 (38.4) |  |  |
  Cycle 13 (Day 168): number analyzed (Participants) | 0 | 0 | 85 | 0 | 0
  Cycle 13 (Day 168) |  |  | 232 (44.1) |  |
  Cycle 12 (Day 231): number analyzed (Participants) | 0 | 3 | 0 | 23 | 26
  Cycle 12 (Day 231) |  | 193 (21.1) |  | 29.3 (34.7) | 173 (38.9)
  Cycle 18 (Day 238): number analyzed (Participants) | 0 | 0 | 3 | 0 | 0
  Cycle 18 (Day 238) |  |  | 171 (27.7) |  |
  Cycle 13 (Day 252): number analyzed (Participants) | 45 | 104 | 0 | 0 | 0
  Cycle 13 (Day 252) | 27.2 (50.4) | 153 (39.6) |  |  |
  Cycle 19 (Day 252): number analyzed (Participants) | 0 | 0 | 65 | 0 | 0
  Cycle 19 (Day 252) |  |  | 253 (37.5) |  |
  Cycle 16 (Day 315): number analyzed (Participants) | 0 | 0 | 0 | 17 | 17
  Cycle 16 (Day 315) |  |  |  | 30.5 (50.6) | 183 (37.8)
  Cycle 24 (Day 322): number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Cycle 24 (Day 322) |  |  | 246 (18.2) |  |
  Cycle 17 (Day 336): number analyzed (Participants) | 37 | 84 | 0 | 0 | 3
  Cycle 17 (Day 336) | 31.4 (48.9) | 168 (48.5) |  |  | 157 (47)
  Cycle 25 (Day 336): number analyzed (Participants) | 0 | 0 | 45 | 0 | 0
  Cycle 25 (Day 336) |  |  | 242 (39.9) |  |
  Cycle 31 (Day 420): number analyzed (Participants) | 0 | 0 | 4 | 0 | 0
  Cycle 31 (Day 420) |  |  | 184 (29.2) |  |
  Cycle 33 (Day 448): number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Cycle 33 (Day 448) |  |  | 80.0 (57.9) |  |
  Cycle 24 (Day 483): number analyzed (Participants) | 0 | 2 | 0 | 8 | 14
  Cycle 24 (Day 483) |  | 152 (7.5) |  | 30.3 (40.1) | 147 (47.0)
  Cycle 25 (Day 504): number analyzed (Participants) | 23 | 57 | 0 | 0 | 0
  Cycle 25 (Day 504) | 29.3 (42.4) | 165 (41.4) |  |  |
  Cycle 37 (Day 504): number analyzed (Participants) | 0 | 0 | 37 | 0 | 0
  Cycle 37 (Day 504) |  |  | 232 (63.8) |  |
  Cycle 32 (Day 651): number analyzed (Participants) | 0 | 0 | 0 | 6 | 12
  Cycle 32 (Day 651) |  |  |  | 23.0 (44.6) | 155 (38.5)
  Cycle 48 (Day 658): number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Cycle 48 (Day 658) |  |  | 169 (25.3) |  |
  Cycle 33 (Day 672): number analyzed (Participants) | 18 | 51 | 0 | 0 | 0
  Cycle 33 (Day 672) | 31.4 (34.0) | 166 (37.7) |  |  |
  Cycle 49 (Day 672): number analyzed (Participants) | 0 | 0 | 27 | 0 | 0
  Cycle 49 (Day 672) |  |  | 255 (42.6) |  |

16. Secondary Outcome: Ctrough of Pembrolizumab in NSCLC Participants (Parts C and F)
Description: Pre-dose samples were collected 24 hours before infusion of pembrolizumab at specified intervals for the determination of Ctrough. Ctrough was defined as the lowest concentration reached by pembrolizumab before the next dose was administered. For the purposes of the Ctrough analysis, samples were collected and analyzed separately for each Part C and F enrolment cohort, and Ctrough was reported for each cohort according to cycle and nominal time after first dose (Day). Results for each cycle reported for arms with N>1 at that timepoint. Ctrough data for solid tumor (Part A) and melanoma (Parts B and D) participants are presented separately and are not included here.
Time Frame: Part C: pre-dose at Cycles 2,5,9,13,17,21 (cycle=21 days); Part F treated every 3 weeks: pre-dose at Cycles 2,3,6,8,12,14,16,24,32 (cycle=21 days); Part F treated every 2 weeks: pre-dose at Cycles 2,3,6,7,8,9,12,16,18,24,32,36,40,48 (cycle=14 days)
Population: All NSCLC participants receiving ≥1 dose of drug and having available samples collected pre-dose before each cycle. Per protocol, Ctrough analyzed separately by Part, dose, and dosing schedule. Due to differing dosing schedules, some time points were not applicable for certain arms (indicated by zero participants analyzed entered in the table).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- NSCLC: Pembrolizumab 10 mg/kg Q3W (Part C); NSCLC: Pembrolizumab 10 mg/kg Q3W (Part F): Participants received pembrolizumab IV at a dose of 10 mg/kg Q3W.
- NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F): Participants received pembrolizumab IV at a dose of 2 mg/kg Q3W.
- NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F): Participants received pembrolizumab IV at a dose of 10 mg/kg Q2W.
Arm/Group | NSCLC: Pembrolizumab 10 mg/kg Q3W (Part C) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Part F)
Number analyzed (Participants) | 33 | 44 | 186 | 230
µg/mL
  Cycle 2 (Day 14): number analyzed (Participants) | 0 | 0 | 186 | 0
  Cycle 2 (Day 14) |  |  | 55.0 (33.8) |
  Cycle 2 (Day 21): number analyzed (Participants) | 33 | 44 | 0 | 230
  Cycle 2 (Day 21) | 52.0 (31.7) | 8.23 (41.1) |  | 43.6 (42.6)
  Cycle 3 (Day 28): number analyzed (Participants) | 0 | 0 | 173 | 0
  Cycle 3 (Day 28) |  |  | 89.3 (39.4) |
  Cycle 3 (Day 42): number analyzed (Participants) | 0 | 39 | 0 | 208
  Cycle 3 (Day 42) |  | 11.8 (62.1) |  | 67.9 (45.5)
  Cycle 4 (Day 42): number analyzed (Participants) | 0 | 0 | 2 | 0
  Cycle 4 (Day 42) |  |  | 173 (36.3) |
  Cycle 6 (Day 70): number analyzed (Participants) | 0 | 0 | 114 | 0
  Cycle 6 (Day 70) |  |  | 149 (40.6) |
  Cycle 5 (Day 84): number analyzed (Participants) | 17 | 0 | 0 | 0
  Cycle 5 (Day 84) | 136 (29.6) |  |  |
  Cycle 7 (Day 84): number analyzed (Participants) | 0 | 0 | 5 | 0
  Cycle 7 (Day 84) |  |  | 159 (19.5) |
  Cycle 8 (Day 98): number analyzed (Participants) | 0 | 0 | 91 | 0
  Cycle 8 (Day 98) |  |  | 180 (42.1) |
  Cycle 6 (Day 105): number analyzed (Participants) | 0 | 28 | 0 | 127
  Cycle 6 (Day 105) |  | 18.3 (40.8) |  | 99.7 (53.9)
  Cycle 9 (Day 112): number analyzed (Participants) | 0 | 0 | 10 | 0
  Cycle 9 (Day 112) |  |  | 145 (44.7) |
  Cycle 8 (Day 147): number analyzed (Participants) | 0 | 21 | 0 | 106
  Cycle 8 (Day 147) |  | 20.6 (46.2) |  | 118 (51.3)
  Cycle 12 (Day 154): number analyzed (Participants) | 0 | 0 | 75 | 0
  Cycle 12 (Day 154) |  |  | 206 (42.6) |
  Cycle 9 (Day 168): number analyzed (Participants) | 8 | 0 | 0 | 2
  Cycle 9 (Day 168) | 168 (26.3) |  |  | 96.8 (47.2)
  Cycle 16 (Day 210): number analyzed (Participants) | 0 | 0 | 33 | 0
  Cycle 16 (Day 210) |  |  | 205 (46) |
  Cycle 12 (Day 231): number analyzed (Participants) | 0 | 14 | 0 | 68
  Cycle 12 (Day 231) |  | 20.0 (60.1) |  | 125 (41.3)
  Cycle 18 (Day 238): number analyzed (Participants) | 0 | 0 | 28 | 0
  Cycle 18 (Day 238) |  |  | 214 (34.7) |
  Cycle 13 (Day 252): number analyzed (Participants) | 9 | 0 | 0 | 0
  Cycle 13 (Day 252) | 197 (47.1) |  |  |
  Cycle 20 (Day 266): number analyzed (Participants) | 0 | 0 | 2 | 0
  Cycle 20 (Day 266) |  |  | 215 (0.98) |
  Cycle 14 (Day 273): number analyzed (Participants) | 0 | 0 | 0 | 4
  Cycle 14 (Day 273) |  |  |  | 121 (56.6)
  Cycle 22 (Day 294): number analyzed (Participants) | 0 | 0 | 3 | 0
  Cycle 22 (Day 294) |  |  | 209 (17.9) |
  Cycle 16 (Day 315): number analyzed (Participants) | 0 | 9 | 0 | 56
  Cycle 16 (Day 315) |  | 23.3 (29.1) |  | 124 (48.6)
  Cycle 24 (Day 322): number analyzed (Participants) | 0 | 0 | 39 | 0
  Cycle 24 (Day 322) |  |  | 234 (33.5) |
  Cycle 17 (Day 336): number analyzed (Participants) | 6 | 0 | 0 | 0
  Cycle 17 (Day 336) | 184 (34.8) |  |  |
  Cycle 26 (Day 350): number analyzed (Participants) | 0 | 0 | 3 | 0
  Cycle 26 (Day 350) |  |  | 202 (13.2) |
  Cycle 18 (Day 357): number analyzed (Participants) | 0 | 0 | 0 | 3
  Cycle 18 (Day 357) |  |  |  | 105 (48.6)
  Cycle 28 (Day 378): number analyzed (Participants) | 0 | 0 | 2 | 0
  Cycle 28 (Day 378) |  |  | 140 (33.5) |
  Cycle 20 (Day 399): number analyzed (Participants) | 0 | 0 | 0 | 2
  Cycle 20 (Day 399) |  |  |  | 81.9 (74.5)
  Cycle 30 (Day 406): number analyzed (Participants) | 0 | 0 | 2 | 0
  Cycle 30 (Day 406) |  |  | 149 (16.2) |
  Cycle 21 (Day 420): number analyzed (Participants) | 6 | 0 | 0 | 0
  Cycle 21 (Day 420) | 167 (40.2) |  |  |
  Cycle 32 (Day 434): number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 32 (Day 434) |  |  | 244 (47.7) |
  Cycle 24 (Day 483): number analyzed (Participants) | 0 | 6 | 0 | 35
  Cycle 24 (Day 483) |  | 24.3 (26) |  | 137 (43.4)
  Cycle 36 (Day 490): number analyzed (Participants) | 0 | 0 | 25 | 0
  Cycle 36 (Day 490) |  |  | 221 (39.9) |
  Cycle 25 (Day 504): number analyzed (Participants) | 2 | 0 | 0 | 0
  Cycle 25 (Day 504) | 207 (67.9) |  |  |
  Cycle 40 (Day 546): number analyzed (Participants) | 0 | 0 | 4 | 0
  Cycle 40 (Day 546) |  |  | 219 (52.2) |
  Cycle 29 (Day 588): number analyzed (Participants) | 3 | 3 | 0 | 0
  Cycle 29 (Day 588) | 173 (39.0) | 32.9 (13.2) |  |
  Cycle 32 (Day 651): number analyzed (Participants) | 0 | 3 | 0 | 25
  Cycle 32 (Day 651) |  | 30.5 (11.6) |  | 141 (49.8)
  Cycle 48 (Day 658): number analyzed (Participants) | 0 | 0 | 21 | 0
  Cycle 48 (Day 658) |  |  | 206 (111.2) |
  Cycle 33 (Day 672): number analyzed (Participants) | 0 | 3 | 0 | 0
  Cycle 33 (Day 672) |  | 40.6 (32.5) |  |

17. Secondary Outcome: Maximum Change From Baseline (CFB) in Tumor Size Assessed by IRC Per RECIST 1.1 According to Programmed Death-Ligand 1 (PD-L1) Immunohistochemical (IHC) Expression Status in Ipilimumab (Ipi)-Exposed and Ipi-Naive Melanoma Participants (Parts B Plus D)
Description: The percent change from baseline in tumor size based on IRC per RECIST 1.1 was reported according to PD-L1 status in Ipi-Exposed and Ipi-Naïve melanoma participants. Tumor PD-L1 status was measured by the tumor proportion score (TPS), which was the percentage of tumor cells identified using IHC analysis that expressed PD-L1. Tumors with ≥1% positive staining for PD-L1 were considered positive. Maximum tumor change was defined as the percent change of the participant's smallest post-baseline tumor size from the baseline. The number of participants in a percent change from baseline range was reported categorically according to PD-L1 status (PD-L1-Positive, PD-L1 Negative, PD-L1 Status Unknown). Negative percent change from baseline values indicate tumor size reduction, with the greatest reduction possible indicated as "≤ -30%". As specified by the protocol, this analysis of melanoma participants was performed according to ipilimumab exposure (Ipi-Exposed and Ipi-Naïve).
Time Frame: Baseline, last available tumor assessment (up to approximately 53 months through Interim Database cut-off date of 18-Sep-2015)
Population: Melanoma participants that received ≥1 dose of study treatment, had a valid PD-L1 expression measurement, and had both baseline and post-baseline tumor assessments. Per protocol, Part A was not analyzed for biomarker analysis. NSCLC (Parts C plus F) participants were analyzed and presented separately and are not included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- MEL (Parts B+D): Ipi-Exposed PD-L1 Positive: Ipi-Exposed melanoma participants that received IV pembrolizumab on study and whose tumors were positive for PD-L1 (TPS ≥1%)
- MEL (Parts B+D): Ipi-Exposed PD-L1 Negative: Ipi-Exposed melanoma participants that received IV pembrolizumab on study and whose tumors were negative for PD-L1 (TPS <1%)
- MEL (Parts B+D): Ipi-Exposed PD-L1 Unknown: Ipi-Exposed melanoma participants that received IV pembrolizumab on study and whose tumors had an unknown PD-L1 status.
- MEL (Parts B+D): All Ipi-Exposed Participants: All Ipi-Exposed melanoma participants that received IV pembrolizumab on study.
- MEL (Parts B+D): Ipi-Naive PD-L1 Positive: Ipi-Naive melanoma participants that received IV pembrolizumab on study and whose tumors were positive for PD-L1 (TPS ≥1%).
- MEL (Parts B+D): Ipi- Naive PD-L1 Negative: Ipi-Naive melanoma participants that received IV pembrolizumab on study and whose tumors were negative for PD-L1 (TPS <1%).
- MEL (Parts B+D): Ipi- Naive PD-L1 Unknown: Ipi-Naive melanoma participants that received IV pembrolizumab on study and whose tumors had an unknown PD-L1 status.
- MEL (Parts B+D): All Ipi- Naive Participants: All Ipi-Naive melanoma participants that received IV pembrolizumab on study.
Arm/Group | MEL (Parts B+D): Ipi-Exposed PD-L1 Positive | MEL (Parts B+D): Ipi-Exposed PD-L1 Negative | MEL (Parts B+D): Ipi-Exposed PD-L1 Unknown | MEL (Parts B+D): All Ipi-Exposed Participants | MEL (Parts B+D): Ipi-Naive PD-L1 Positive | MEL (Parts B+D): Ipi- Naive PD-L1 Negative | MEL (Parts B+D): Ipi- Naive PD-L1 Unknown | MEL (Parts B+D): All Ipi- Naive Participants
Number analyzed (Participants) | 176 | 37 | 47 | 260 | 140 | 50 | 61 | 251
Participants
  Number of Participants with ≤ -30% CFB | 93 | 8 | 25 | 126 | 94 | 22 | 35 | 151
  Number of Participants with > -30% to <20% CFB | 57 | 17 | 14 | 88 | 32 | 10 | 11 | 53
  Number of Participants with ≥ 20% CFB | 26 | 12 | 8 | 46 | 14 | 18 | 15 | 47

18. Secondary Outcome: Maximum Change From Baseline (CFB) in Tumor Size Assessed by IRC Per RECIST 1.1 According to PD-L1 IHC Expression Status in Prior Treatment (TRT)-Naïve and Previously-Treated NSCLC Participants (Parts C Plus F)
Description: Percent CFB in tumor size based on IRC per RECIST 1.1 was reported according to PD-L1 status in prior treatment-naïve and previously-treated NSCLC participants. Tumor PD-L1 status was measured by TPS, which was the percentage of tumor cells identified using IHC analysis that expressed PD-L1, as follows: TPS ≥50% =tumor strongly positive, TPS of 1%-49% =tumor weakly positive, TPS <1% =tumor considered negative, or TPS unknown. Maximum tumor change for a participant was defined as the percent change of the participant's smallest post-baseline tumor size from baseline. The number of participants in a percent CFB range was reported categorically according to PD-L1 status (TPS ≥50%, TPS = 1-49%, TPS <1%, TPS Unknown). Negative percent CFB values indicate tumor size reduction, with the greatest reduction possible indicated as "≤ -30%". As specified by the protocol, analysis of NSCLC participants was performed according to prior treatment exposure (Treatment Naive and Previously Treated).
Time Frame: as for outcome 17
Population: NSCLC participants that received ≥1 dose of study treatment, had a valid PD-L1 expression measurement, and had both baseline and post-baseline tumor assessments. Per protocol, Part A was not analyzed for biomarker analysis. Melanoma (Parts B plus D) participants were analyzed and presented separately and are not included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- NSCLC (Parts C+F): TRT-Naïve TPS ≥50%: Prior treatment (TRT)-naïve NSCLC participants that received IV pembrolizumab on study and whose tumors were strongly positive for PD-L1 (TPS ≥50%).
- NSCLC (Parts C+F): TRT-Naïve TPS = 1-49%: Prior TRT-naïve NSCLC participants that received IV pembrolizumab on study and whose tumors were weakly positive for PD-L1 (TPS 1-49%).
- NSCLC (Parts C+F): TRT-Naïve TPS <1%: Prior TRT-naïve NSCLC participants that received IV pembrolizumab on study and whose tumors were negative for PD-L1 (TPS <1%).
- NSCLC (Parts C+F): TRT-Naïve TPS Unknown: Prior TRT-naïve NSCLC participants that received IV pembrolizumab on study and whose tumors had an unknown PD-L1 status.
- NSCLC (Parts C+F): All TRT-Naïve Participants: All prior TRT-naïve NSCLC participants that received IV pembrolizumab on study.
- NSCLC (Parts C+F): Previously Treated TPS ≥50%: Previously-treated NSCLC participants that received IV pembrolizumab on study and whose tumors were strongly positive for PD-L1 (TPS ≥50%).
- NSCLC (Parts C+F): Previously Treated TPS = 1-49%: Previously-treated NSCLC participants that received IV pembrolizumab on study and whose tumors were weakly positive for PD-L1 (TPS 1-49%).
- NSCLC (Parts C+F): Previously Treated TPS <1%: Previously-treated NSCLC participants that received IV pembrolizumab on study and whose tumors were negative for PD-L1 (TPS <1%).
- NSCLC (Parts C+F): Previously Treated TPS Unknown: Previously-treated NSCLC participants that received IV pembrolizumab on study and whose tumors had an unknown PD-L1 status.
- NSCLC (Parts C+F): All Previously Treated Participants: All Previously-treated NSCLC participants that received IV pembrolizumab on study.
Arm/Group | NSCLC (Parts C+F): TRT-Naïve TPS ≥50% | NSCLC (Parts C+F): TRT-Naïve TPS = 1-49% | NSCLC (Parts C+F): TRT-Naïve TPS <1% | NSCLC (Parts C+F): TRT-Naïve TPS Unknown | NSCLC (Parts C+F): All TRT-Naïve Participants | NSCLC (Parts C+F): Previously Treated TPS ≥50% | NSCLC (Parts C+F): Previously Treated TPS = 1-49% | NSCLC (Parts C+F): Previously Treated TPS <1% | NSCLC (Parts C+F): Previously Treated TPS Unknown | NSCLC (Parts C+F): All Previously Treated Participants
Number analyzed (Participants) | 23 | 39 | 10 | 9 | 81 | 110 | 137 | 66 | 38 | 351
Participants
  Number of Participants with ≤ -30% CFB | 16 | 15 | 2 | 4 | 37 | 58 | 42 | 15 | 14 | 129
  Number of Participants with > -30% to <20% CFB | 7 | 20 | 6 | 4 | 37 | 32 | 65 | 38 | 14 | 149
  Number of Participants with ≥ 20% CFB | 0 | 4 | 2 | 1 | 7 | 20 | 30 | 13 | 10 | 73

19. Secondary Outcome: Disease Control Rate (DCR) According to RECIST 1.1 as Assessed by IRO in Melanoma Participants (Parts B and D)
Description: DCR was defined as the percentage of participants who had a CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of diameters of target lesions), or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD]). The percentage of participants who experienced a confirmed CR, PR, or SD according to RECIST 1.1 as assessed by IRO was reported as the DCR for each melanoma dose arm (Parts B plus D).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 162 | 313 | 180 | 0 | 0 | 0
Percentage of Participants |  |  |  |  |  |  | 48.1 [40.2 to 56.1] | 47.6 [42.0 to 53.3] | 56.1 [48.5 to 63.5] |  |  |

20. Secondary Outcome: Duration of Response (DOR) According to RECIST 1.1 as Assessed by IRO in Melanoma Participants (Parts B and D)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. DOR assessments were based on IRO with confirmation. The DOR according to RECIST 1.1 for all participants who experienced a confirmed CR or PR was reported for each melanoma dose arm (Parts B plus D).
Time Frame: From time of first documented evidence of CR or PR through Interim Database cut-off date of 18-Sep-2015 (Up to approximately 53 months)
Population: All melanoma (Parts B plus D) participants that received ≥1 dose of study treatment and who demonstrated a confirmed response (CR or PR). Per protocol, Part A (dose-escalation) was not analyzed for efficacy. NSCLC (Parts C plus F) participants were analyzed and presented separately and are not included in this analysis.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 92 | 66 | 0 | 0 | 0
Weeks |  |  |  |  |  |  | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment) | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment) | NA [16.1 to NA] — NA=Median DOR and DOR range upper limit not reached (no progressive disease by time of last disease assessment) |  |  |

21. Secondary Outcome: Progression Free Survival (PFS) According to RECIST 1.1 as Assessed by IRO in Melanoma Participants (Parts B Plus D)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS according to RECIST 1.1 as assessed by IRO was reported for each melanoma dose arm (Parts B plus D).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 162 | 313 | 180 | 0 | 0 | 0
Months |  |  |  |  |  |  | 4.9 [2.8 to 8.3] | 3.7 [2.8 to 5.5] | 5.6 [3.3 to 10.0] |  |  |

22. Secondary Outcome: Overall Survival (OS) in Melanoma Participants (Parts B Plus D)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. OS was reported for each melanoma dose arm (Parts B plus D).
Time Frame: Up to approximately 91 months (through Final Database cut-off date of 05-Nov-2018)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 162 | 313 | 180 | 0 | 0 | 0
Months |  |  |  |  |  |  | 23.1 [17.8 to 33.1] | 22.5 [18.5 to 32.0] | 26.8 [19.6 to 41.8] |  |  |

23. Secondary Outcome: DCR According to irRC as Assessed by Investigator in Melanoma Participants (Parts B Plus D)
Description: DCR according to irRC was defined as the percentage of participants who had a irCR (complete disappearance of all tumor lesions whether measurable or not, and no new lesions), irPR (decrease in SPD of ≥50% by a consecutive assessment ≥4 weeks after first documentation), or SD (neither sufficient shrinkage to qualify for irPR nor sufficient increase to qualify for PD [at least a 25% increase in SPD relative to nadir (minimum recorded tumor burden) with confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented]). The percentage of participants who experienced a confirmed CR, PR, or SD according to irRC as assessed by the investigator was reported as the DCR for each melanoma dose arm (Parts B plus D).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 162 | 313 | 180 | 0 | 0 | 0
Percentage of Participants |  |  |  |  |  |  | 62.3 [54.4 to 69.8] | 62.6 [57.0 to 68.0] | 69.4 [62.2 to 76.1] |  |  |

24. Secondary Outcome: DOR According to irRC as Assessed by Investigator in Melanoma Participants (Parts B Plus D)
Description: For participants who demonstrated a confirmed irCR (complete disappearance of all tumor lesions whether measurable or not, and no new lesions) or irPR (decrease in SPD of ≥50% by a consecutive assessment ≥4 weeks after first documentation) according to irRC, DOR was defined as the time from first documented evidence of an irCR or irPR until PD or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. According to irRC, PD was defined as at least a 25% increase in SPD relative to nadir (minimum recorded tumor burden) with confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented. The DOR according to irRC as assessed by the investigator for all participants who experienced a confirmed irCR or irPR was reported for each melanoma dose arm (Parts B plus D).
Time Frame: From time of first documented evidence of iCR or iPR through Interim Database cut-off date of 18-Sep-2015 (Up to approximately 53 months)
Population: All melanoma (Parts B plus D) participants that received ≥1 dose of study treatment and who demonstrated a confirmed irRC response (irCR or irPR). Per protocol, Part A (dose-escalation) was not analyzed for efficacy. NSCLC (Parts C plus F) participants were analyzed and presented separately and are not included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 57 | 125 | 82 | 0 | 0 | 0
Months |  |  |  |  |  |  | NA [2.1 to NA] — NA=Median DOR and DOR range upper limit not reached (no progressive disease by time of last disease assessment) | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment) | NA [2.7 to NA] — NA=Median DOR and DOR range upper limit not reached (no progressive disease by time of last disease assessment) |  |  |

25. Secondary Outcome: PFS According to irRC as Assessed by Investigator in Melanoma Participants (Parts B Plus D)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. According to irRC, PD was defined as at least a 25% increase in SPD relative to nadir (minimum recorded tumor burden) with confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented. PFS according to irRC as assessed by the investigator was reported for each melanoma dose arm (Parts B plus D).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 162 | 313 | 180 | 0 | 0 | 0
Months |  |  |  |  |  |  | 8.2 [5.6 to 13.6] | 6.6 [5.5 to 10.5] | 9.6 [5.6 to 19.3] |  |  |

26. Secondary Outcome: DCR According to RECIST 1.1 as Assessed by IRC in NSCLC Participants (Parts C Plus F)
Description: DCR was defined as the percentage of participants who had a CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of diameters of target lesions), or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD]). The percentage of participants who experienced a confirmed CR, PR, or SD according to RECIST 1.1 as assessed by IRC was reported as the DCR for each NSCLC dose arm (Parts C plus F).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 287 | 202
Percentage of Participants |  |  |  |  |  |  |  |  |  | 50.8 [37.7 to 63.9] | 51.6 [45.6 to 57.5] | 49.0 [41.9 to 56.1]

27. Secondary Outcome: DOR According to RECIST 1.1 as Assessed by IRC in NSCLC Participants (Parts C Plus F)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until PD or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. DOR assessments were based on IRC with confirmation. The DOR according to RECIST 1.1 for all participants who experienced a confirmed CR or PR was reported for each NSCLC dose arm (Parts C plus F).
Time Frame: as for outcome 20
Population: All NSCLC (Parts C plus F) participants that received ≥1 dose of study treatment and who demonstrated a confirmed response (CR or PR). Per protocol, Part A (dose-escalation) was not analyzed for efficacy. Melanoma (Parts B and D) participants were analyzed and presented separately and are not included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 62 | 39
Months |  |  |  |  |  |  |  |  |  | NA [NA to 19.0] — NA=Median DOR and DOR range lower limit not reached (no progressive disease by time of last disease assessment) | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment) | 20.7 [2.8 to NA] — NA=DOR range upper limit not reached (no progressive disease by time of last disease assessment)

28. Secondary Outcome: PFS According to RECIST 1.1 as Assessed by IRC in NSCLC Participants (Parts C Plus F)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS according to RECIST 1.1 as assessed by IRC was reported for each NSCLC dose arm (Parts C plus F).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 287 | 202
Months |  |  |  |  |  |  |  |  |  | 3.3 [2.0 to 4.4] | 3.7 [2.4 to 4.2] | 3.4 [2.3 to 4.2]

29. Secondary Outcome: OS in NSCLC Participants (Parts C Plus F)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. OS was reported for each NSCLC dose arm (Parts C plus F).
Time Frame: Up to approximately 91 months (through Final Database cut-off date of 05-Nov-2018)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 287 | 202
Months |  |  |  |  |  |  |  |  |  | 8.9 [5.8 to 15.4] | 13.1 [10.3 to 17.3] | 13.4 [9.4 to 15.7]

30. Secondary Outcome: DCR According to irRC as Assessed by Investigator in NSCLC Participants (Parts C Plus F)
Description: DCR according to irRC was defined as the percentage of participants who had a irCR (complete disappearance of all tumor lesions whether measurable or not, and no new lesions), irPR (decrease in SPD of ≥50% by a consecutive assessment ≥4 weeks after first documentation), or SD (neither sufficient shrinkage to qualify for irPR nor sufficient increase to qualify for PD [at least a 25% increase in SPD relative to nadir (minimum recorded tumor burden) with confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented]). The percentage of participants who experienced a confirmed CR, PR, or SD according to irRC as assessed by the investigator was reported as the DCR for each NSCLC dose arm (Parts C plus F).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 287 | 202
Percentage of Participants |  |  |  |  |  |  |  |  |  | 57.4 [44.1 to 70.1] | 62.7 [56.8 to 68.3] | 65.3 [58.3 to 71.9]

31. Secondary Outcome: DOR According to irRC as Assessed by Investigator in NSCLC Participants (Parts C Plus F)
Description: For participants who demonstrated a confirmed irCR (complete disappearance of all tumor lesions whether measurable or not, and no new lesions) or irPR (decrease in SPD of ≥50% by a consecutive assessment ≥4 weeks after first documentation) according to irRC, DOR was defined as the time from first documented evidence of an irCR or irPR until PD or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. According to irRC, PD was defined as at least a 25% increase in SPD relative to nadir (minimum recorded tumor burden) with confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented. The DOR according to irRC as assessed by the investigator for all participants who experienced a confirmed irCR or irPR was reported for each NSCLC dose arm (Parts C plus F).
Time Frame: as for outcome 24
Population: as for outcome 27
Measure: Median (Full Range); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 83 | 45
Months |  |  |  |  |  |  |  |  |  | NA [NA to 21.9] — NA= Median DOR and DOR range lower limit not reached (no progressive disease by time of last disease assessment) | NA [NA to NA] — NA= Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment) | NA [3.0 to NA] — NA=Median DOR and DOR range upper limit not reached (no progressive disease by time of last disease assessment)

32. Secondary Outcome: PFS According to irRC as Assessed by Investigator in NSCLC Participants (Parts C Plus F)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. According to irRC, PD was defined as at least a 25% increase in SPD relative to nadir (minimum recorded tumor burden) with confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented. PFS according to irRC as assessed by the investigator was reported for each NSCLC dose arm (Parts C plus F).
Time Frame: Up to approximately 53 months (through Interim Database cut-off date of 18-Sep-2015)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 287 | 202
Months |  |  |  |  |  |  |  |  |  | 4.3 [2.3 to 6.1] | 4.4 [4.0 to 6.2] | 5.6 [4.1 to 6.5]

ADVERSE EVENTS:
Time Frame: Up to approximately 91 months (through Final Database cut-off date of 05-Nov-2018)
Description: All-Cause Mortality reported for all randomized/enrolled participants. AEs reported for All Treated Population.Per protocol, disease progression on study not considered an AE unless related to drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to drug excluded as AEs. 5 participants were not assessed by cutoff and were followed to study completion; end of study assessments are missing for these 5 and status is unknown
Groups:
- Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2): During Cycle 1 participants received pembrolizumab dose titration from 0.005 mg/kg to 0.3 mg/kg to 2.0 mg/kg on Days 1, 8, and 22, administered as an IV infusion over 30 minutes. Participants received 2 mg/kg Q3W starting with Cycle 2.
Arm/Group | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F)
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/3 | 6/12 | 2/4 | 1/3 | 5/6 | 111/164 | 213/321 | 110/183 | 52/61 | 240/296 | 166/203
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/3 | 3/10 | 0/4 | 2/3 | 2/6 | 69/162 | 129/313 | 79/180 | 34/61 | 119/287 | 86/202
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 8/10 | 4/4 | 3/3 | 5/6 | 158/162 | 303/313 | 175/180 | 55/61 | 271/287 | 191/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) (N=4) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) (N=3) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) (N=10) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) (N=4) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) (N=3) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) (N=6) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) (N=162) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) (N=313) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) (N=180) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) (N=61) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) (N=287) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F) (N=202)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 6 (6) | 2 (2) | 2 (2) | 2 (3) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecalith (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 3 (3) | 0 (0) | 6 (7) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 3 (3) | 3 (3) | 6 (6) | 2 (3)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bacillus bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 8 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 9 (12) | 8 (8) | 6 (8) | 7 (8) | 13 (15)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound decomposition (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical observation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 4 (8) | 0 (0) | 2 (2) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insulin resistant diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (11) | 8 (14) | 4 (4) | 0 (0) | 2 (3) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 10 (13) | 7 (8) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 7 (7) | 2 (2) | 2 (2) | 9 (9) | 5 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 5 (5) | 2 (2) | 3 (3) | 14 (19) | 8 (9)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 2 (3) | 2 (3) | 7 (8) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 4 (4) | 2 (2) | 8 (9) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 6 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated cryptococcosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Listeriosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis listeria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumors: Pembrolizumab 1 mg/kg Q2W (Part A) (N=4) | Solid Tumors: Pembrolizumab 3 mg/kg Q2W (Part A) (N=3) | Solid Tumors: Pembrolizumab 10 mg/kg Q2W (Parts A+A1) (N=10) | Solid Tumors: Pembrolizumab Titration Cohort 1 Q3W (Part A2) (N=4) | Solid Tumors: Pembrolizumab Titration Cohort 2 Q3W (Part A2) (N=3) | Solid Tumors: Pembrolizumab Titration Cohort 3 Q3W (Part A2) (N=6) | MEL: Pembrolizumab 2 mg/kg Q3W (Parts B+D) (N=162) | MEL: Pembrolizumab 10 mg/kg Q3W (Parts B+D) (N=313) | MEL: Pembrolizumab 10 mg/kg Q2W (Part B) (N=180) | NSCLC: Pembrolizumab 2 mg/kg Q3W (Part F) (N=61) | NSCLC: Pembrolizumab 10 mg/kg Q3W (Parts C+F) (N=287) | NSCLC: Pembrolizumab 10 mg/kg Q2W (Part F) (N=202)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 27 (58) | 61 (113) | 30 (57) | 5 (5) | 37 (52) | 38 (72)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 3 (3) | 0 (0) | 4 (5) | 5 (5)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 16 (17) | 23 (25) | 28 (37) | 6 (7) | 20 (26) | 22 (22)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 9 (10) | 10 (12) | 0 (0) | 2 (2) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 6 (6) | 21 (22) | 10 (11) | 2 (2) | 7 (8) | 3 (3)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 13 (13) | 7 (11) | 0 (0) | 4 (5) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 10 (11) | 10 (10) | 0 (0) | 10 (10) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 26 (40) | 38 (49) | 31 (55) | 5 (5) | 29 (37) | 20 (24)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 22 (22) | 13 (18) | 1 (1) | 10 (12) | 6 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 45 (60) | 68 (85) | 41 (65) | 10 (12) | 47 (51) | 46 (56)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 54 (112) | 111 (195) | 70 (145) | 12 (16) | 67 (127) | 39 (62)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 23 (23) | 18 (22) | 3 (4) | 12 (16) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 11 (13) | 11 (14) | 0 (0) | 7 (7) | 5 (5)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (22) | 10 (12) | 13 (19) | 1 (2) | 17 (17) | 5 (5)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (2) | 2 (3) | 56 (91) | 108 (144) | 69 (109) | 9 (11) | 60 (79) | 47 (60)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 2 (2) | 0 (0) | 5 (6) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 5 (6) | 4 (6) | 3 (3) | 7 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 33 (50) | 62 (84) | 43 (56) | 9 (13) | 44 (59) | 28 (53)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 20 (41) | 50 (82) | 28 (72) | 7 (11) | 24 (44) | 23 (46)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 19 (23) | 12 (18) | 2 (4) | 22 (23) | 20 (24)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 17 (18) | 43 (60) | 24 (28) | 0 (0) | 12 (12) | 12 (12)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (4)
Fatigue (General disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (2) | 2 (2) | 3 (4) | 77 (157) | 163 (249) | 106 (220) | 17 (23) | 122 (172) | 78 (110)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 10 (10) | 3 (4) | 0 (0) | 2 (2) | 3 (3)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 25 (27) | 11 (21) | 1 (2) | 5 (5) | 4 (6)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 28 (35) | 53 (68) | 37 (48) | 4 (4) | 38 (47) | 23 (27)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (11) | 14 (17) | 11 (17) | 5 (9) | 24 (27) | 20 (26)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 16 (24) | 50 (72) | 38 (53) | 5 (9) | 36 (63) | 24 (29)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 8 (9) | 7 (8) | 4 (4) | 7 (9) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 10 (12) | 7 (23)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 4 (4) | 5 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 26 (43) | 31 (45) | 26 (47) | 4 (6) | 8 (11) | 3 (4)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 4 (4) | 8 (9)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 2 (3) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 8 (9) | 7 (7) | 4 (4) | 18 (22) | 11 (11)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 9 (14) | 4 (6) | 1 (1) | 7 (7) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 13 (16) | 19 (26) | 0 (0) | 7 (11) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 23 (49) | 28 (47) | 28 (48) | 1 (1) | 34 (66) | 25 (32)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 16 (18) | 25 (43) | 20 (37) | 2 (2) | 16 (21) | 11 (26)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 12 (14) | 11 (11) | 2 (2) | 2 (2) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (12) | 10 (20) | 9 (12) | 2 (2) | 10 (12) | 10 (12)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (17) | 30 (38) | 21 (30) | 2 (3) | 16 (23) | 11 (19)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 33 (53) | 23 (36) | 1 (2) | 21 (25) | 13 (20)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 16 (21) | 13 (21) | 5 (7) | 14 (17) | 9 (14)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 16 (33) | 5 (5) | 1 (1) | 9 (19) | 8 (10)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (10) | 14 (16) | 13 (19) | 3 (4) | 12 (17) | 6 (9)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 16 (21) | 36 (53) | 13 (15) | 4 (6) | 26 (32) | 23 (25)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (20) | 17 (44) | 8 (22) | 0 (0) | 8 (11) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 36 (47) | 70 (92) | 47 (59) | 10 (14) | 88 (125) | 55 (62)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (17) | 13 (19) | 10 (12) | 1 (1) | 14 (16) | 6 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 19 (60) | 11 (42) | 2 (3) | 23 (41) | 16 (50)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 17 (48) | 12 (25) | 0 (0) | 8 (15) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 17 (37) | 13 (26) | 4 (5) | 13 (13) | 7 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 15 (24) | 16 (24) | 3 (3) | 17 (22) | 12 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 20 (38) | 10 (17) | 2 (2) | 16 (17) | 13 (18)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 18 (30) | 22 (36) | 3 (6) | 16 (28) | 16 (26)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (16) | 15 (29) | 8 (15) | 0 (0) | 10 (14) | 5 (8)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 50 (103) | 93 (175) | 60 (128) | 9 (18) | 54 (89) | 47 (82)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 35 (47) | 53 (74) | 32 (43) | 5 (6) | 36 (47) | 28 (38)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 7 (10) | 18 (19) | 5 (5) | 0 (0) | 5 (6) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (15) | 13 (16) | 14 (17) | 3 (4) | 10 (11) | 7 (20)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 16 (22) | 19 (20) | 15 (21) | 1 (1) | 11 (12) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 17 (20) | 11 (12) | 0 (0) | 21 (30) | 13 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (20) | 29 (33) | 17 (21) | 7 (9) | 24 (29) | 17 (23)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 9 (9) | 7 (11) | 0 (0) | 3 (3) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 23 (38) | 48 (68) | 45 (85) | 2 (2) | 23 (35) | 24 (28)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 16 (18) | 5 (5) | 3 (3) | 6 (8) | 11 (14)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 30 (45) | 40 (58) | 32 (47) | 2 (2) | 21 (29) | 12 (15)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 2 (2) | 7 (10) | 6 (9) | 1 (2) | 6 (7) | 4 (10)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 21 (34) | 34 (46) | 26 (34) | 5 (7) | 40 (52) | 20 (24)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 11 (15) | 6 (6) | 0 (0) | 11 (11) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 36 (58) | 79 (127) | 52 (91) | 5 (7) | 41 (46) | 19 (23)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (12) | 9 (10) | 9 (11) | 1 (1) | 4 (4) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 5 (5) | 5 (6) | 0 (0) | 3 (3) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (16) | 14 (19) | 13 (22) | 1 (1) | 14 (16) | 4 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 19 (22) | 13 (15) | 3 (3) | 7 (9) | 9 (13)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (10) | 2 (2) | 1 (1) | 3 (4) | 4 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 24 (27) | 15 (17) | 4 (7) | 17 (17) | 12 (12)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 9 (9) | 12 (13) | 1 (1) | 7 (8) | 14 (14)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 29 (39) | 36 (41) | 19 (24) | 3 (5) | 32 (34) | 16 (16)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 51 (81) | 92 (151) | 58 (92) | 10 (13) | 86 (127) | 51 (72)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 30 (44) | 65 (85) | 42 (60) | 10 (14) | 80 (97) | 52 (66)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (12) | 10 (13) | 9 (9) | 2 (2) | 19 (20) | 10 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (7) | 1 (1) | 2 (4) | 21 (24) | 15 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (19) | 27 (42) | 18 (24) | 0 (0) | 11 (14) | 9 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (12) | 23 (33) | 14 (26) | 0 (0) | 12 (13) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 4 (4) | 3 (4) | 6 (9) | 15 (16) | 15 (17)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 12 (17) | 10 (14) | 2 (3) | 12 (16) | 5 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (21) | 20 (30) | 12 (15) | 3 (3) | 20 (24) | 22 (27)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 9 (10) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 27 (32) | 12 (15) | 3 (3) | 19 (24) | 21 (25)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (13) | 18 (22) | 10 (12) | 0 (0) | 10 (12) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 8 (8) | 10 (10) | 0 (0) | 5 (5) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 15 (20) | 18 (23) | 15 (16) | 0 (0) | 2 (2) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 49 (92) | 99 (165) | 66 (121) | 4 (7) | 52 (73) | 27 (36)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 9 (9) | 7 (9) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 47 (84) | 87 (189) | 45 (103) | 7 (10) | 43 (71) | 27 (42)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 22 (37) | 6 (8) | 0 (0) | 9 (11) | 8 (12)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 21 (33) | 44 (57) | 28 (37) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 6 (7) | 5 (5) | 0 (0) | 6 (7) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 31 (87) | 11 (21) | 2 (2) | 11 (19) | 8 (11)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 16 (21) | 5 (5) | 0 (0) | 5 (6) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 16 (19) | 9 (16) | 1 (1) | 6 (12) | 6 (23)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 13 (16) | 5 (5) | 1 (1) | 8 (9) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT01295827/Prot_SAP_000.pdf